CLINICAL TRIAL: NCT07365917
Title: Effect of Lumbar Core Stabilization Exercises on Craniovertebral Angle and Functional Outcome in Patients With Cervical Radiculopathy
Brief Title: Effect of Core Stabilization Exercises on Patients With Cervical Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Gamal Abdelbasset, Demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/006086
Record Dates: First submitted 2026-01-13; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cervical Radiculopathy
Keywords: Core stabilization exercises; craniovertebral angle
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator)
  Interventions: Other: conventional physical therapy program
- study group (Experimental)
  Interventions: Other: Core stabilization exercises; Other: conventional physical therapy program

INTERVENTIONS:
Other: Core stabilization exercises — participants in study group will receive 30 mins and 3 sessions per week for 4 weeks
  Arms: study group
Other: conventional physical therapy program — conventional physical therapy program will include TENS, hot pack, US, manual therapy and strengthening exercises

SUMMARY:
The goal of this clinical trial is to evaluate the effect of core stabilization exercise on functional outcome and craniovertebral angle which is the angle of forward head , in adults with cervical radiculopathy. The main questions it aims to answer are:

* Is there a significant effect of core stabilization exercises (CSEs) on craniovertebral angle (CVA) in patients with cervical radiculopathy?
* Is there a significant effect of core stabilization exercises (CSEs) on functional outcome in patients with cervical radiculopathy? Researchers will compare effect of adding core stabilization exercises to conventional physical therapy program (TENS, hot pack, US, manual therapy and strengthening exercises) Vs conventional physical therapy program alone to see if there is a beneficial effect of adding core stabilization exercises to physical therapy program Participants in study group will perform core stabilization exercises in addition to conventional PT program while participants in control group will receive conventional PT program

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Posterolateral cervical disc proplapse at level of C5-C6 and C6-C7 levels
2. Neck Disability Index (NDI) score exceeding 20%.
3. Neck pain of mild to moderate intensity (VAS ≥ 3).
4. Their symptoms lasting for a duration exceeding six weeks
5. Three out of four elements are positive in the following tests: spurling test, distraction test, upper limb tension test, shoulder abduction test.
6. Body mass index should not exceed 30 kg/m².
7. Patients complaining from neck pain and unilateral radicular pain, parathesia, motor manifestations or hyporeflexia
8. Their age will range from 35 to 50 years.
9. Their craniovertebral angle is less than 49 degrees.
10. Their mean of cervical joint position error is larger than 4.5 degrees.

Exclusion Criteria:

1. Cervical mylopathy or spinal tumors
2. History of cervical spine surgeries
3. Cervical fractures
4. Vertebrobasilar insufficiency (VBI)
5. Bone Infection

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Craniovertebral Angle | from enrollment to the end of treatment at 4 weeks
  Craniovertebral angle ( CVA ) will be measured through lateral photography of patients. Before capturing the picture, Plastic markers will be placed on C7 vertebra and on tragus of ear. Then the picture will be uploaded to kinovea software to measure CVA by measuring the angle between a line connecting two plastic markers and the horizontal. Values more than 49 degrees are considered abnormal indicating forward head posture while values lower than 49 degrees indicate normal head position
Arabic Version of Neck Disability Index (NDI) | from enrollment to the end of treatment at 4 weeks
  Functional outcome will be assessed though Arabic Version of Neck Disability Index (NDI) which is a 10-item self-reported questionnaire. It measures the influence of neck pain on functioning and disability. The patient will be informed that this questionnaire had been designed to give us how your pain had affected your ability to function in daily life. Personal care, lifting, reading, work, driving, sleeping, recreational activities, pain intensity, concentration, and headache are examples of these questions. Each question is assessed on a six-point scale ranging from 0 (no disability) to 5 (major disability). The score will be calculated by adding the scores of each item together. The overall score is out of 50. The results can be expressed as a percentage by multiplying the score by two. The higher NDI score, the greater patient's perceived disability due to neck pain. The Arabic version of NDI is a strong valid method for assessing self-rated disability in patients with neck pain

SECONDARY OUTCOMES:
Neck Pain | from enrollment to the end of treatment at 4 weeks
  Neck pain will be assessed though Visual Analogue Scale (VAS) which is used to measure the severity of neck pain. It is a straight line with one end representing no pain and the other end representing the worst imaginable pain. The subject will mark a point on the line that corresponds to the current level of pain he or she experiences. Higher values indicate higher levels of pain while lower values indicate lower levels of pain
Cervical Proprioception | from enrollment to the end of treatment at 4 weeks
  Cervical proprioception will be assessed through measurement of cervical Joint Position Error (JPE). Instruments that will be utilized are laser pointer device mounted on participant's head and a chart with a reference point at its center. the chart is positioned 90cm in front of patients. A test of repositioning to a neutral head position (NHP) will be carried out to determine JPE. Participants will move their head away from the start position at the center of the chart which is the NHP to full range and then attempt to reposition the head back to the starting point as accurately as possible while they are blindfolded. The difference between the starting position (zero) and the returning point in the plane of movement will be measured in centimeters and then converted to degrees using this formula angle = tan-1 [error distance/90 cm]. Normal cervical JPE is 4.5 degree. Higher values indicate poor cervical proprioception

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Egypt